CLINICAL TRIAL: NCT00106977
Title: Clinical Study of Muenke Syndrome (FGFR3-Related Craniosynostosis)
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050131; 05-HG-0131
Record Dates: First submitted 2005-04-01; First posted 2005-04-04 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Craniosynostosis; Muenke Syndrome
Keywords: Coronal Craniosynostosis; Hearing Loss; Pro250 Arg Mutation; Tarsal Coalition; Carpal Coalition; Muenke Syndrome; Craniosynostosis
MeSH Terms: conditions — Craniosynostoses; Muenke Syndrome; Hearing Loss; Tarsal Coalition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Family: Family members (typically parents or siblings) of probands with Muenke syndrome are alsoeligible to participate.
- Patient: Subjects who have had confirmation of a p. Pro250Arg mutation in FGFR3 by a CLIA-certified laboratory.

SUMMARY:
This study will explore the range and type of medical and developmental problems in patients with Muenke syndrome, a condition that results when one or more of the suture between the bones of the skull close before birth. Because of the premature closure, the skull is not able to grow in its natural shape; instead, it compensates with growth in areas of the skull where the sutures have not yet closed. This can result in an abnormally shaped head, wide-set eyes, and flattened cheekbones. Patients may also have an enlarged head, abnormalities of the hands or feet, and hearing loss.

The fibroblast growth factor receptor 3 (FGFR3) gene, which is involved in the development and maintenance of bone tissue, plays a role in Muenke syndrome. In some cases, the FGFR3 mutation is inherited from a parent with Muenke syndrome; in other cases, where there is no family history of the disorder, the mutation occurs anew. A better understanding of this gene may lead researchers to develop better treatments and genetic counseling for people affected by Muenke syndrome.

Patients with Muenke syndrome and their blood relatives may be eligible for this study. Family members with confirmed Muenke syndrome will have genetic counseling, and patients undergo the following tests and procedures:

* Review of medical records and test results.
* Questionnaires about the patient's prenatal, birth, newborn, and past medical history; family history; growth and development; medications; and current therapies.
* Physical, neurological, ear, nose and throat, dental, and eye examinations.
* Neuropsychological testing to assess cognitive thinking abilities.
* Hearing evaluation. This includes an audiology test in which the patients listens to soft tones through earphones; a power reflectance test in which a chirping sound is heard through an earpiece placed at the entrance to the ear canal, and possibly an ABR/ASSR test, in which electrodes are attached to the forehead, earlobes, and behind the ears to measure brain waves in response to certain conditions.
* MRI scan of the brain. MRI uses a strong magnetic field and radio waves to produce detailed pictures of the brain. During the scan, the patient lies on a table in a narrow cylinder (the scanner), wearing ear plugs to muffle loud noises that occur with electrical switching of the magnetic fields.
* MRI scan of the middle and inner ear. This test is similar to the MRI, but uses a dye injected in a vein to enhance the images.
* CT scan of the skull. CT uses x-rays to produce 3-dimensional images of the part of the body studied.
* Dental evaluation with x-rays.
* Skeletal survey (x-rays of all bones of the body).
* Developmental assessment of IQ testing.
* Blood tests for research purposes. A cell line may be established for use in future research.
* Medical photographs to demonstrate clinical features, including side and front views of the face, head, and other parts of the body that may be involved in Muenke syndrome, like the hands and feet.
* Other consultations or tests as clinically indicated

DETAILED DESCRIPTION:
Craniosynostosis is a common craniofacial abnormality caused by premature fusion of one or several sutures of the skull. The prevalence of craniosynostosis is approximately 1 in 2,100 to 3,000 births. Originally described by our group, Muenke syndrome (OMIM # 602849) is a specific form of craniosynostosis caused by a single nucleotide transversion in fibroblast growth factor receptor 3 (FGFR3), c.749C>G, resulting in p.Pro250Arg. Individuals carrying the defining mutation variably manifest coronal suture craniosynostosis, developmental delay, deafness, and carpal and tarsal bone fusion. The purpose of the present study is to increase our understanding of the clinical manifestations of Muenke syndrome through detailed physical, developmental, neurologic, dental, ophthalmologic, otolaryngologic, audiologic, radiologic, and genetic/genomic studies. We also plan to examine the spectrum of clinical characteristics of Muenke syndrome to facilitate early diagnosis and clinical management, including genetic counseling. To accomplish this, we plan to enroll approximately 10-20 probands, as well as their family members each year, with an enrollment ceiling of 200 probands. Our study has three arms. The clinical arm is the major focus of our study. Patients and their families will be seen at the NIH Clinical Center and Children's National Medical Center. Individuals with Muenke syndrome who are unable or unwilling to come to the NIH, can submit their medical records, including a copy of the molecular testing, for review. The second arm is genetic/genomic studies with the goal of investigating modifying factors that relate to disease severity and expression. The third arm consists of a cognitive function, development and hearing questionnaire to be completed by patients online, via phone or mail.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects who have had confirmation of a Pro250Arg mutation in FGFR3 by a CLIA-certified laboratory. Our research team must receive a photocopy of the positive test result in order to enroll a patient in the study. All races and genders are known to be at risk for Muenke syndrome. Nationality or place of origin is not a specific barrier to participation.

Family members (typically parents or siblings) of probands with Muenke syndrome are also eligible to participate.

* Since the penetrance of Muenke syndrome is incomplete, any at risk individual will be given the option of enrolling in the research study for FGFR3 testing. Those individuals who are found to carry the p.Pro250Arg mutation may benefit from interventions like hearing screening or speech evaluations that would alter their medical management. Variable expressivity is another characteristic of Muenke syndrome and carrier status and adequate genetic counseling are important. Individuals with the mutation will be invited to participate in the clinical and/or medical record review arms of the study
* Unaffected family members of a proband enrolled in the clinical protocol may choose to provide a blood sample and/or participate in the behavioral arm of the study. These information will be used only for purposes of further research on Muenke syndrome.

Patient of interest cases. Geneticists and genetic counselors may refer individuals who are suspected to have Muenke syndrome, but who have not yet been tested for the FGFR3 Pro250Arg mutation. The purpose of enrolling these subjects is to evaluate a wider spectrum of patients for the mutation causing Muenke syndrome. Testing for the Pro250Arg mutation maybe performed at the discretion of our research group. Those individuals who are found to carry the Pro250 Arg mutation may be invited to participate in the study. Individuals who do not carry the mutation but that have an affected first degree family member will be invited to participate in the

genomic and/or survey arm of the study.

EXCLUSION CRITERIA:

* Anyone unwilling to provide informed consent (for themselves as adults, or on behalf of their children as minors) or assent.
* We reserve the right to exclude individuals for whom the medical risks of travel and evaluation at NIH appear to outweigh the benefits of study participation.

Description and justification of inclusion/exclusion of participants. (age, gender, ethnicity, prisoners, pregnant women, fetuses, decisionally-impaired, healthy volunteers, lab personnel)

It is our intention to remove as many economic, cultural, geographic, racial, and gender barriers as we reasonably can to promote participation of individuals with Muenke syndrome and their families for research purposes. The study will include pediatric and decisionally-impaired individuals, because these characteristics are possible with Muenke syndrome. Pregnant or nursing women may be limited in their participation in some aspects of the study.

As described above, Muenke syndrome has been demonstrated to occur in persons of different ethnic backgrounds. We would make every reasonable effort to encourage the enrollment and participation of a wide spectrum of individuals.

-Pregnant women will not be excluded.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have had confirmation of a p.Pro250Arg mutation in FGFR3 by a CLIA-certified laboratory. Family members (typically parents or siblings) of probands with Muenke syndrome are also eligible to participate.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2005-03-31 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Understanding | Ongoing
  The objective of this study is primarily to increase our understanding of the genetics and clinical characteristics of Muenke syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Kruszka, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Bellus GA, Gaudenz K, Zackai EH, Clarke LA, Szabo J, Francomano CA, Muenke M. Identical mutations in three different fibroblast growth factor receptor genes in autosomal dominant craniosynostosis syndromes. Nat Genet. 1996 Oct;14(2):174-6. doi: 10.1038/ng1096-174. PMID 8841188
- [Background] Muenke M, Gripp KW, McDonald-McGinn DM, Gaudenz K, Whitaker LA, Bartlett SP, Markowitz RI, Robin NH, Nwokoro N, Mulvihill JJ, Losken HW, Mulliken JB, Guttmacher AE, Wilroy RS, Clarke LA, Hollway G, Ades LC, Haan EA, Mulley JC, Cohen MM Jr, Bellus GA, Francomano CA, Moloney DM, Wall SA, Wilkie AO, et al. A unique point mutation in the fibroblast growth factor receptor 3 gene (FGFR3) defines a new craniosynostosis syndrome. Am J Hum Genet. 1997 Mar;60(3):555-64. PMID 9042914
- [Background] Moloney DM, Wall SA, Ashworth GJ, Oldridge M, Glass IA, Francomano CA, Muenke M, Wilkie AO. Prevalence of Pro250Arg mutation of fibroblast growth factor receptor 3 in coronal craniosynostosis. Lancet. 1997 Apr 12;349(9058):1059-62. doi: 10.1016/s0140-6736(96)09082-4. PMID 9107244
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2005-HG-0131.html